CLINICAL TRIAL: NCT03401840
Title: A Multicenter Prospective Phase II Study of Postoperative Hypofractionated Stereotactic Body Radiotherapy (SBRT) in the Treatment of Early Stage Oropharyngeal and Oral Cavity Cancers With High Risk Margins.
Brief Title: STEREO-POSTOP 01 (PostOperative Hypofractionated Stereotactic Body Radiotherapy ) - GORTEC 2017-03
Acronym: STEREOPOSTOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Collaborators: GORTEC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-A02058-45; PHRC-K16-164 (Other Grant/Funding Number: Directorate of Health Care Supply (DGOS), National Cancer Institute (INCa), France)
Record Dates: First submitted 2017-12-19; First posted 2018-01-17 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Neoplasms
Keywords: Head and neck cancers; Radiation oncology; Stereotactic radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- postoperative SBRT (Experimental): SBRT consists of a total dose of 36 Gy in 6 fractions over 11-13 days
  Interventions: Radiation: postoperative hypofractionated stereotactic radiotherapy

INTERVENTIONS:
Radiation: postoperative hypofractionated stereotactic radiotherapy — total dose of 36Gy in 6 fractions over 11-13 days

SUMMARY:
The main objective of this national, open-label, non-randomized phase II trial is to evaluate severe late toxicity of postoperative hypofractionated stereotactic radiotherapy (SBRT) in the treatment of early stage oropharyngeal and oral cavity cancer with high risk margins.

ELIGIBILITY:
Inclusion Criteria:

* Operated squamous cell carcinoma of oral cavity (lips excepted) or oropharynx
* pT1 or pT2 ((UICC 7th edition 2009)
* Indication of postoperative tumor site irradiation (retained in multidisciplinary tumor board) with at least one of the following criteria :

  * positive R1 margin (re-resection not proposed)
  * close margin < 5 mm (re-resection not proposed)
  * Margin estimated at risk, with uncertain pathological margin (re-resection not proposed)
* N0 after surgical management of the neck (neck dissection or sentinel lymph node biopsy) or pN1 without extracapsular extension (carcinological neck dissection)
* Age ≥ 18 years
* ECOG status ≤ 2
* Written signed informed consent before any specific procedure of the protocol
* Affiliation to a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Other histology than squamous cell carcinoma
* pT3 or pT4
* pT2>3cm and R1 with concurrent chemoradiotherapy decided in multidisciplinary tumor board
* Lymphovascular invasion justifying neck irradiation
* Neck irradiation decided in multidisciplinary tumor board
* Lack of at least one of the following elements :

  * pre-operative medical imaging (CT scan or MRI)
  * endoscopy report
  * surgery report
  * pathological report
* Prior radiotherapy to the head and neck area
* Distant metastasis
* Pregnant or nursing (lactating) woman
* women or men of childbearing age not taking adequate contraceptive measure
* participation in another investigational study within 4 weeks prior to inclusion
* History of other malignancy within 5 years prior enrollment except for basal cell carcinoma of the skin or carcinoma in situ of the cervix
* Persons deprived of their liberty, under guardianship or curatorship, or unable to follow the trial for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
severe late toxicity | from 3 months to 2 years following the end of radiotherapy
  2-year toxicity of grade ≥ 3 related to SBRT according to CTCAE V4.03 classification.

SECONDARY OUTCOMES:
Local control | 2 years following the end of radiotherapy
  2-year local control rate - Any local recurrence (T) will be considered as an event.
Locoregional control | 2 years following the end of radiotherapy
  2-year locoregional control rate - Any local (T) or lymph node (N) recurrence will be considered as an event
Acute toxicity | from the first fraction to 3 months after the end of radiotherapy
  ≤ 3-month toxicity of grade ≥ 3 related to SBRT according to CTCAE V4.03 classification.
disease free survival (DFS) | 2 years following the end of radiotherapy
  2-year DFS rate - DFS is time from randomization to the date of first occurrence of any locoregional recurrence, distant progression or death from any cause.
Overall survival (OS) | 2 years following the end of radiotherapy
  2-year OS rate - OS is defined as time from randomization to death from any cause
Quality of life (global evaluation) | at baseline, 1 month, 1 year and 2 years post radiotherapy
  evaluated by EORTC QLQC30
Quality of life (specific evaluation for Head and Neck Cancer) | at baseline, 1 month, 1 year and 2 years post radiotherapy
  evaluated by EORTC QLQ HN35 module
Nutritional impact | during 2 years following the end of radiotherapy
  evaluated by weight loss
Nutritional support | during 2 years following the end of radiotherapy
  evaluated by the use of feeding tubes
Predictive factors of toxicity | 2 years following the end of radiotherapy
  clinical and/or dosimetric factors associated to late severe toxicities (grade ≥ 3 related to SBRT according to CTCAE V4.03 classification).

CONTACTS AND LOCATIONS:
Overall Officials: Julian BIAU, Principal Investigator — Centre Jean Perrin
Locations (24):
- France (24):
  - Institut Sainte Catherine, Avignon
  - Institut Bergonié, Bordeaux
  - Polyclinique bordeaux Nord Aquitaine, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier de Bretagne Sud /Site du Scorff, Lorient
  - Centre Léon Bérard, Lyon
  - Hôpital Nord Franche-Comté, Montbéliard
  - Institut de Cancérologie de Montpellier, Val d'Aurelle, Montpellier
  - Hôpital Tenon, Paris
  - Hôpital Universitaire Pitié Salpêtrière - Charles Foix, Paris
  - Hôpital Haut-Lévêque - Groupe hospitalier sud - CHU de Bordeaux, Pessac
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Institut Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier Privé Saint Grégoire, Saint-Grégoire
  - Institut de Cancérologie de l'ouest, Site René Gauducheau, Saint-Herblain
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - Clinique Pasteur, Toulouse
  - Institut Claudius Regaud, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biau J, Sun X, Liem X, Faivre JC, Eker E, Blanchard P, Tao Y, Dore M, Maingon P, Vulquin N, Alfonsi M, Thureau S, Huguet F, Racadot S, Thivat E, Molnar I, Boisselier P, Guihard S, Gallocher O, Dupin C, Batard S, Bourhis J, Lapeyre M. Postoperative SBRT and Severe Late Toxic Effects in Early-Stage Oropharyngeal and Oral Cavity Cancers: The STEREOPOSTOP-GORTEC 2017-03 Nonrandomized Clinical Trial. JAMA Netw Open. 2025 Dec 1;8(12):e2549975. doi: 10.1001/jamanetworkopen.2025.49975. PMID 41632122
- [Derived] Biau J, Thivat E, Millardet C, Saroul N, Pham-Dang N, Molnar I, Pereira B, Durando X, Bourhis J, Lapeyre M. A multicenter prospective phase II study of postoperative hypofractionated stereotactic body radiotherapy (SBRT) in the treatment of early-stage oropharyngeal and oral cavity cancers with high risk margins: the STEREO POSTOP GORTEC 2017-03 trial. BMC Cancer. 2020 Aug 5;20(1):730. doi: 10.1186/s12885-020-07231-3. PMID 32758188